CLINICAL TRIAL: NCT00632619
Title: A Novel Multimodal Intervention for Children With ADHD and Impaired Mood
Brief Title: Group-Based Behavioral Therapy Combined With Stimulant Medication for Treating Children With Attention Deficit Hyperactivity Disorder and Impaired Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH080791 (NIH); R34MH080791 (NIH); DDTR B2-NDH
Record Dates: First submitted 2008-03-07; First posted 2008-03-11 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Subthreshold Manic States in Children; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive stimulant medication therapy and referrals to community-based psychosocial treatments.
  Interventions: Drug: Stimulant medication therapy; Behavioral: Community-based psychosocial treatment
- 2 (Experimental): Participants will receive stimulant medication therapy and group-based behavior therapy.
  Interventions: Behavioral: Group-based behavior therapy; Drug: Stimulant medication therapy

INTERVENTIONS:
Behavioral: Group-based behavior therapy — Group-based behavior therapy with a parenting class will include 12 weeks of sessions that focus on reducing oppositional and aggressive behaviors. Children will participate in 12 weeks of social skills training integrated with a cognitive behavioral therapy (CBT) component to target mood symptoms. Parents will learn ways to identify and address their child's mood problems, communicate better with their child, and work with school staff to address academic and behavioral problems.
  Arms: 2
Drug: Stimulant medication therapy — All participants will be stabilized on an FDA-approved stimulant medication for 2 to 6 weeks prior to therapy assignment.
Behavioral: Community-based psychosocial treatment — Participants will receive referrals to community-based psychosocial treatments that will focus on ADHD symptoms and management of aggression.
  Arms: 1

SUMMARY:
This study will evaluate the effectiveness of an integrative group psychosocial therapy combined with stimulant medication in treating children with attention deficit hyperactivity disorder plus impairments in mood.

DETAILED DESCRIPTION:
There has been increasing recognition that many children with attention deficit hyperactivity disorder (ADHD) exhibit depressive and manic-like symptoms suggestive of major depressive disorder (MDD) and bipolar disorder (BP). Many children with ADHD plus impairments in mood display symptoms of irritability, affective instability, and reactive aggression, but they typically lack the hallmark symptoms, such as extreme mood cycles and sustained depressed mood, that lead to a BD or MDD diagnosis. Significant debate exists as to whether these children have a true comorbid mood disorder, making treatment of mood symptoms in ADHD children controversial. ADHD is traditionally treated with stimulant medications and/or behavior modification therapy. However, little is known about the safety of stimulants in ADHD children with manic symptoms. Also, no treatments exist that are designed to simultaneously improve both ADHD and mood problems in children. Psychosocial treatments hold particular promise for ADHD children with impairments in mood because they are well-studied pediatric treatments with little risk of worsening mood symptoms. This study will develop an integrative psychosocial treatment that includes aspects of cognitive behavioral therapy (CBT) and psychoeducational techniques for pediatric and adult mood disorders. The study will then evaluate the effectiveness of the integrative psychosocial treatment, called group behavior therapy, combined with stimulant medication in improving moods and enhancing treatment responses in children with ADHD and impairments in mood.

Participation in the study will last between 5 and 6 months. All eligible participants will begin treatment with stimulant medications for 2 to 6 weeks, or until an optimal medication dosage has been determined. During this medication dosing phase, study staff will collect weekly ratings of the child participant's behavior at home and school, and participants will be seen weekly by study doctors to monitor medication dosage. Upon achieving an optimal dose, child participants will answer questions about their mood and behavior.

Participants who are still exhibiting mood problems will then be assigned randomly to receive 12 weeks of either group behavior therapy or community-based psychosocial treatment, while still continuing on their prescribed medications. Group behavior therapy sessions for child participants will focus on improving mood and ability to maintain friendships, practicing ways to better control emotions, and learning effective problem solving skills. Child participants will also be given weekly homework assignments to practice learned therapy skills. Group behavior therapy sessions for parent participants will teach parents ways to identify and address their child's mood problems, communicate better with their child, and work with school staff to address academic and behavioral problems. Participants assigned to community-based psychosocial treatment will not receive any counseling services as part of the study, but they will be referred to community services.

Every 6 weeks during the therapy phase, all participants will answer repeat questions about their mood and behavior. Six weeks after completing the therapy phase, participants will return for a final follow-up visit, which will include repeat questions, rating of the child participant's mood and symptoms, and meeting with a study doctor to check medications.

ELIGIBILITY:
Inclusion Criteria:

* ADHD combined subtype with evidence of depressive or manic-like symptoms, as assessed by CDRS, YMRS, and Washington University in St. Louis Kiddie Schedule for Affective Disorders and Schizophrenia, that persist after stimulant treatment

Exclusion Criteria:

* Full Scale IQ less than 80
* Current seizure disorder or history of seizures requiring treatment or other significant neurological problems
* History of other medical problems for which stimulant treatment may involve considerable risk, including cardiac arrhythmias, hypertension, Tourette's disorder, or history of severe tic exacerbations caused by stimulant exposure (Note: child with uncomplicated tic disorders or a family history of tic disorders will not be excluded as stimulants are well tolerated in a majority of such cases)
* Meets full criteria for Type I or II bipolar disorder or any child manifesting mood symptoms (manic or depressive), such as significant suicidal ideation or psychotic symptoms that require emergent pharmacological treatment or hospitalization
* History or concurrent diagnosis of any of the following disorders: pervasive developmental disorder, schizophrenia or other psychotic disorders, post-traumatic stress disorder, sexual disorders, organic mental disorder, or eating disorder
* No longer manifests impairing manic/depressive symptoms after stimulant therapy based on CDRS-R greater than 27 or YMRS greater than 11 with Clinical Global Impressions-Severity 3 or greater

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James G. Waxmonsky, MD, Principal Investigator — Florida International University
Locations (1):
- Center for Children and Families at Florida International University, Miami, Florida, United States

REFERENCES:
- [Derived] Waxmonsky JG, Waschbusch DA, Belin P, Li T, Babocsai L, Humphery H, Pariseau ME, Babinski DE, Hoffman MT, Haak JL, Mazzant JR, Fabiano GA, Pettit JW, Fallahazad N, Pelham WE. A Randomized Clinical Trial of an Integrative Group Therapy for Children With Severe Mood Dysregulation. J Am Acad Child Adolesc Psychiatry. 2016 Mar;55(3):196-207. doi: 10.1016/j.jaac.2015.12.011. Epub 2015 Dec 28. PMID 26903253
- See also: Click here for more information on this study at the Center for Children and Families at State University of New York at Buffalo — http://casgroup.fiu.edu/ccf/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited as two cohorts- 50% in each wave. Wave one was recruited in Buffalo NY in the summer of 2009, from referrals from local pediatricians and therapists and mailings to families. The study was then moved to Florida International University where the second cohort was recruited from 9/10 to 12/10 using similar procedures.
Pre-assignment Details: Subjects were assessed at intake on the current ADHD medication regimen to make sure that they needed additional treatment beyond what they were currently receiving. There was no washout prior to enrollment.
Groups:
- Medication and Community Treatment Group: Participants will receive stimulant medication therapy and referrals to community-based psychosocial treatments.
  Stimulant medication therapy : All participants will be stabilized on an FDA-approved stimulant medication for 4 to 8 weeks prior to therapy assignment.
  Community-based psychosocial treatment : Participants will receive referrals to community-based psychosocial treatments that will focus on ADHD symptoms and management of aggression.
- Medication and Novel Therapy Group: Participants will receive stimulant medication therapy and group-based behavior therapy.
  Stimulant medication therapy : All participants will be stabilized on an FDA-approved stimulant medication for 4 to 8 weeks prior to therapy assignment.
  Group-based behavior therapy : Group-based behavior therapy with a parenting class will include 12 weeks of sessions that focus on reducing oppositional and aggressive behaviors. Children will participate in 12 weeks of social skills training integrated with a cognitive behavioral therapy (CBT) component to target mood symptoms. Parents will learn ways to identify and address their child's mood problems, communicate better with their child, and work with school staff to address academic and behavioral problems.
Period: Overall Study
Arm/Group | Medication and Community Treatment Group | Medication and Novel Therapy Group
Started | 33 (first cohort started 9/11/09 second cohort started 12/7/11) | 35 (first cohort started 9/11/09 second cohort started 12/7/11)
Completed | 25 (1. st cohort completed follow up by 5/24/10 2. nd cohort completed follow up 7/18/11) | 31 (1. st cohort completed follow up by 5/24/10 2. nd cohort completed follow up 7/18/11)
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medication and Community Treatment Group | Medication and Novel Therapy Group | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 35 | 68
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.4 (1.5) | 9.3 (1.6) | 9.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 26 | 24 | 50
Region of Enrollment [Number; unit: participants]
  United States | 33 | 35 | 68

OUTCOME MEASURES:

1. Secondary Outcome: Young Mania Rating Scale (YMRS) Score
Description: rates manic like symptoms in children; 7 items ranging from 0-4 and 4 items on a 0-8 scale; higher scores indicate more severe symptom severity (min total score=0, max=60). There are no subscales. Symptom severity information is obtained from direct interview of parent and child. It was initially selected as the primary outcome but prior to commencement of data collection the Mood Severity Index (MSI) was chosen instead based on recently published work in a related study (see above).
Time Frame: Measured at weeks 12 (endpoint)
Population: all subjects who were successfully stabilized on stimulant medication and then entered therapy phase; subjects not able to tolerate stimulant med for ADHD or whose mood symptoms resolved with optimization of their stimulant dose were not included in the therapy phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication and Community Treatment Group | Medication and Novel Therapy Group
Number analyzed (Participants) | 25 | 31
units on a scale | 10.08 (4.65) | 8.58 (5.05)
Statistical Analysis 1: Comparison: Medication and Community Treatment Group vs Medication and Novel Therapy Group; A 2 x 2 repeated measures analysis (with time as within-subject factor and group as between-subject factor) was performed to compare the two groups on this measure at two time points (i.e., baseline at week 0 and endpoint at week 12) and infer treatment success accordingly. The null hypothesis signified that there would be no difference between the groups over time, thus, there would be no difference in treatments. Statistical power was calculated as Cohen's d; Test type: Superiority or Other; p = 0.106, ANOVA

2. Primary Outcome: Mood Severity Index Measures Severity of Mood Symptoms (MSI).Range of 0-116; Clinicians Give to Parents and Child to Get Composite Score; Higher Scores=Greater Severity; 0-10=no Symptoms, 11-20=Mild Symptoms, 21to 35 =Moderate Symptoms and >35 is Severe
Description: averaged Composite of endpoint ratings from the Children's Depression Rating Scale (CDRS used to measure depressive symptoms) and Young mania rating scale (MRS used to measure manic like symptoms) that has been used before as primary outcome in treatment studies of children with a mixture of affective symptoms (Fristad, et al., 2009). Prior to commencement of data collection, we elected to use it as the primary mood measure for the therapy phase of the trial over the initially selected YMRS as subjects either had to have elevations on the YMRS or CDRS but not necessarily both to be eligible. Hence, some subjects had very low YMRS scores at baseline which is why we chose the MSI over the YMRS.
Time Frame: measured at week 12 (endpoint)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication and Community Treatment Group | Medication and Novel Therapy Group
Number analyzed (Participants) | 25 | 31
units on a scale | 17.33 (7.29) | 13.82 (6.03)
Statistical Analysis 1: Comparison: Medication and Community Treatment Group vs Medication and Novel Therapy Group; A 2 x 2 repeated measures analysis (with time as within-subject factor and group as between-subject factor) was performed to compare the two groups on this measure at two time points (i.e., baseline which was week 0 and endpoint at week 12) and infer treatment success accordingly. The null hypothesis signified that there would be no difference between the groups over time, thus, there would be no difference in treatments. Statistical power was calculated as Cohen's d; Test type: Superiority or Other; p = 0.015, ANOVA

3. Secondary Outcome: Disruptive Behavior Disorder Scale Score for ADHD Symptoms
Description: sum of severity rating for all 18 DSM (Diagnostic and Statistics Manual for Mental Disorders) IV ADHD symptoms and two from DSM 3R on a 0 to 3 scale obtained from parent rating; range is from 0 to 60 with higher numbers indicating more severe symptoms
Time Frame: Measured at Week12 (endpoint)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication and Community Treatment Group | Medication and Novel Therapy Group
Number analyzed (Participants) | 25 | 31
units on a scale | 25.5 (10.94) | 25.10 (9.12)
Statistical Analysis 1: Comparison: Medication and Community Treatment Group vs Medication and Novel Therapy Group; A 2 x 2 repeated measures analysis (with time as within-subject factor and group as between-subject factor) was conducted to compare the two groups on this measure at two time points (i.e., baseline at week 0 and endpoint at week 12) and infer treatment success accordingly. The null hypothesis signified that there would be no difference between the groups over time, thus, there would be no difference in treatments. Statistical power was calculated as Cohen's d; Test type: Superiority or Other; p = 0.38, ANOVA

4. Secondary Outcome: Children's Depression Rating Scale-Revised (CDRS-R) Total Score
Description: rates 17 items of depression on a severity scale using information obtained from parent and child. Higher numbers indicate more severity symptoms and range is from 17 to 113.
Time Frame: Measured at Week 12 (endpoint)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication and Community Treatment Group | Medication and Novel Therapy Group
Number analyzed (Participants) | 25 | 31
units on a scale | 28.20 (6.46) | 25.10 (3.96)
Statistical Analysis 1: Comparison: Medication and Community Treatment Group vs Medication and Novel Therapy Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.016, ANOVA

5. Secondary Outcome: Disruptive Behavior Disorder Scale Score for ODD Symptoms
Description: parents rating all DSM symptoms of Oppositional Defiant Disorder on a 0-3 severity scale with higher scores indicating more severe symptoms and range is from 0-27 (8 DSM IV items and I item from DSM 3R)
Time Frame: week 12 (endpoint)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication and Community Treatment Group | Medication and Novel Therapy Group
Number analyzed (Participants) | 25 | 31
units on a scale | 11.13 (6.22) | 10.31 (4.73)
Statistical Analysis 1: Comparison: Medication and Community Treatment Group vs Medication and Novel Therapy Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.095, ANOVA

ADVERSE EVENTS:
Time Frame: for two years- from first subject enrolling in summer of 2009 to last follow up assessment done summer of 2011. Three controls dropped prior to any study treatments so they are not included in the adverse event analysis which is why the N is 30 not 33.
Description: Pittsburgh side effect rating scale given at every assessment point to assess medication related side effects. It lists 13 common (appetite loss, insomnia) and rare (hallucinations) adverse events associated with stimulants on a 0-3 likert with 3 being severe.
  The suicide item from the CDRS was used to systematically measure suicidal ideation.
Arm/Group | Medication and Community Treatment Group | Medication and Novel Therapy Group
Serious Adverse Events (participants affected / at risk) | 1/30 | 4/35
Other Adverse Events (participants affected / at risk) | 16/30 | 20/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication and Community Treatment Group (N=30) | Medication and Novel Therapy Group (N=35)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — subject was admitted to hospital due to worsening of asthma. The child was discharged the next day at baseline health. Therapy treatment had ended 3 weeks prior but participant was on study medication which was deemed unrelated to the event.
threat of self injurious behavior (Psychiatric disorders) | 1 (1) | 0 (0) — Control who became upset at school when asked to do work and picked up scissors and threatened(but did not attempt) to cut his hand. He was sent for emergency psychiatric assessment. He was discharged home that day at his baseline mental status.
appendix removed (Gastrointestinal disorders) | 0 (0) | 1 (1) — Therapy subject hospitalized for appendicitis. he had appendix removed and discharged home 48hrs later with no sequelae.
aggression towards other (Psychiatric disorders) | 0 (0) | 1 (1) — Therapy subject with history of aggression who became physically aggressive towards another student and then a teacher. She was hospitalized for 48hrs. No psychotropic medication was started and she was discharged at baseline mental status.
expresssed suicial ideation (Psychiatric disorders) | 0 (0) | 1 (1) — Therapy subject who expressed suicidal ideation at school but made no attempt. He was hospitalized, diagnosed with pervasive developmental disorder traits & anxiety disorder. He was started on exclusionary medication so was discontinued from study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication and Community Treatment Group (N=30) | Medication and Novel Therapy Group (N=35)
worried/anxious (Psychiatric disorders) | 3 (3) | 6 (6) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant
picking at skin, fingers, nails, lips (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant
repetitive movements/motor tics (Nervous system disorders) | 1 (1) | 3 (3) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant
dull/tired (General disorders) | 2 (2) | 1 (1) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant
stomachaches (Gastrointestinal disorders) | 1 (1) | 2 (2) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant
crabby or irritable (Psychiatric disorders) | 5 (5) | 9 (9) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant
loss of appetite (General disorders) | 5 (5) | 6 (6) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant
insomnia (General disorders) | 3 (3) | 6 (6) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant
tearful/sad affect (Psychiatric disorders) | 2 (2) | 1 (1) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant.
dull or tired looking (Psychiatric disorders) | 2 (2) | 1 (1) — measured on the Pittsburgh Side effect rating scale which lists the most common (as well as rare ) adverse events seen with stimulant medications; each is rated on 0-3 with 0-none 3= severe. items rated 2 or more are considered clinically relevant

LIMITATIONS AND CAVEATS:
relatively small sample size, the lack of a gold standard measurement for mood dysregulation in children, run at a specialty mental health research center and therapy subjects had more contact with study staff which may have impacted results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No